CLINICAL TRIAL: NCT03084289
Title: A Phase I Study to Assess the Safety and Immunogenicity of Novel Routes of Administration of Plasmodium Falciparum Malaria Vaccine Candidates ChAd63 and MVA Encoding ME-TRAP.
Brief Title: A Study to Assess the Safety and Immunogenicity of a Candidate Malaria Vaccine Using Novel Routes of Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC064
Record Dates: First submitted 2017-03-03; First posted 2017-03-20 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-08

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group 1 (Experimental): Group 1 will receive ChAd63-METRAP at the dose of 5x10^8 vp i.v.
  Interventions: Biological: ChAd63-METRAP
- Group 2 (Experimental): Group 2 will receive ChAd63-METRAP at the dose of 5x10^9 vp i.v.
  Interventions: Biological: ChAd63-METRAP
- Group 3 (Experimental): Group 3 will receive ChAd63-METRAP at the dose of 5x10^10 vp i.v.
  Interventions: Biological: ChAd63-METRAP
- Group 4 (Experimental): Group 4 will receive ChAd63-METRAP at the dose of 5x10^10 vp s.c.
  Interventions: Biological: ChAd63-METRAP
- Group 5 (Experimental): Group 5 will receive ChAd63-METRAP at the dose of 2x10^11 vp s.c.
  Interventions: Biological: ChAd63-METRAP
- Group 6 (Experimental): Group 6 will receive MVA METRAP at the dose of 2 x 10^6 pfu i.v.
  Interventions: Biological: MVA ME-TRAP
- Group 7 (Experimental): Group 7 will receive MVA METRAP at the dose of 2 x 10^7 pfu i.v.
  Interventions: Biological: MVA ME-TRAP
- Group 8 (Experimental): Group 8 will receive MVA METRAP at the dose of 2 x 10^8 pfu i.v.
  Interventions: Biological: MVA ME-TRAP

INTERVENTIONS:
Biological: ChAd63-METRAP — The candidate vaccine applicable to the clinical trial is the Chimpanzee adenovirus 63 expressing Multiple epitopes and thrombospondin related adhesion protein.
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5
Biological: MVA ME-TRAP — The candidate vaccine applicable to the clinical trial is the Modified Vaccinia virus Ankara expressing Multiple epitopes and thrombospondin related adhesion protein.
  Arms: Group 6; Group 7; Group 8

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of novel routes of administration of the candidate malaria vaccines ChAd63 encoding ME-TRAP and MVA encoding ME-TRAP.

30-33 Healthy adult volunteers will be recruited in Oxford.

All vaccinations will be administered intravenously or subcutaneously. Each volunteer will receive a single vaccination of ChAd63 ME-TRAP or MVA ME-TRAP at different doses depending on the group.

DETAILED DESCRIPTION:
Group1 consists of 3 volunteers receiving i.v. ChAd63 ME-TRAP at the dose of 5x10^8 vp.

Group 2 consists of 3 volunteers receiving i.v. ChAd63 ME-TRAP at the dose of 5x10^9 vp.

Group 3 consists of 9 volunteers receiving i.v. ChAd63 ME-TRAP at the dose of 5x10^10vp.

Group 4 consists of 3 volunteers receiving s.c. ChAd63 ME-TRAP at the dose of 5x10^10 vp.

Group 5 consists of 3 volunteers receiving s.c. ChAd63 ME-TRAP at the dose of 2x10^11 vp.

Group 6 consists of 3 volunteers receiving i.v. MVA ME-TRAP at the dose of 2x10^6 pfu.

Group 7 consists of 3 volunteers receiving i.v. MVA ME-TRAP at the dose of 2x10^7 pfu.

Group 8 consists of 3-6 volunteers receiving i.v. MVA ME-TRAP at the dose of 2x10^8 pfu.

The first Group 1 volunteer to receive intravenous ChAd63 ME-TRAP will be vaccinated alone. Safety data for the first 72 hours following vaccination must be satisfactorily reviewed before the remaining group 1 volunteers are vaccinated. The safety data for the first 72 hours following vaccination for all the volunteers in the group will again be reviewed before the first volunteer in the higher dose group 2 is vaccinated. Safety data for the first 72 hours following vaccination of this volunteer must be satisfactorily reviewed before the remaining group 2 volunteers are vaccinated. Similarly the safety data for the first 72 hours following vaccination for all the volunteers in this group will again be reviewed before the first volunteer in the higher dose group 3 is vaccinated. Once there is satisfactory review of the safety data of the first 72 hours post vaccination for this volunteer, the remaining group 3 volunteers will be enrolled to receive IV vaccination.

An identical process will be followed for the enrolment of groups 6 - 8 receiving MVA ME-TRAP intravenously. Once three group 8 volunteers have received vaccination and there has been a satisfactory safety review at 72 hours, the chief investigator will make a decision as to whether or not to enrol the final three volunteers on the basis of the immunology data - and whether further determination of immunogenicity is needed.

In parallel with Group 1, the first Group 4 volunteer to receive subcutaneous Chad63 ME-TRAP will be vaccinated alone. Safety data for the first 72 hours following vaccination must be satisfactorily reviewed before the remaining group 4 volunteers are vaccinated. The safety data for the first 72 hours following vaccination for all the volunteers in the group will again be reviewed before the first volunteer in the higher dose group 5 is vaccinated. Once there is satisfactory review of the safety data of the first 72 hours post vaccination for this volunteer, the remaining group 5 volunteers will be enrolled to receive SC vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis in relation to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition likely to affect participation in the study
* Bleeding disorder (e.g. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* History of clinical malaria (any species)
* Travel to a malaria endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry, coagulation, haematology blood tests or urinalysis
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Incidence of occurrence of emergent adverse events related to subcutaneous and intravenous administration of ChAd63 ME-TRAP and MVA ME-TRAP in healthy malaria-naïve volunteers | 3 months
  The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events (including solicited local or systemic reactogenicity signs and symptoms for 7 days following the vaccination; occurrence of unsolicited adverse events for 28 days following vaccination, and the occurrence of serious adverse events throughout the 3 month study duration).

SECONDARY OUTCOMES:
Identify potential biomarkers of vaccine deposition in the liver (biomolecules measured will include: liver enzymes and plasma cytokine levels). | 3 months
  Changes in potential biomarkers before and after vaccination will be assessed to identify markers biologically consistent with hepatocyte perturbation and inflammation. Some of the methodology will include: clotting assays (e.g. D-dimer levels), peripheral blood gene transcriptional profiling and some exploratory proteomic analysis of urine and plasma.
Assess changes in immune response before and after vaccination using exploratory immunological assays. | 3 months
  Measures of immunogenicity generated in malaria naïve individuals of subcutaneous and intravenous administration of ChAd63 ME-TRAP, may include: ELISPOT (to enumerate IFN-γ producing T cells), flow cytometry and intracellular cytokine staining (to enumerate and functionally characterise immune cell populations such as T cells (e.g. CD4+ and CD8+) and B cells) and possibly gene expression profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V Hill, DPhill FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No